CLINICAL TRIAL: NCT04967989
Title: Clarifying the Optimal Application of SLT Therapy Trial
Acronym: COAST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Eye Institute (NEI) (NIH); West Virginia University (Other)
Responsible Party: Principal Investigator, Balasubramani Goundappa, Research Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21060171; UG1EY031651 (NIH); UG1EY031654 (NIH); STUDY21080018 (Other: University of Pittsburgh)
Record Dates: First submitted 2021-06-27; First posted 2021-07-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma and Ocular Hypertension
Keywords: glaucoma; selective laser trabeculoplasty; clinical trial
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: The COAST trial underwent a design modification in response to a planned interim analysis. The original and current designs are described here.
  Initial Design: Subjects are randomized at study entry to initial SLT at standard or low energy. Subjects who reach Month 12 without discontinuing study treatment are randomized a second time to annual low-energy repeat SLT or as-needed standard energy repeat SLT. There are 2 arms in the first 12 months of the study and 2 arms in Months 13-48.
  Current deign: Subjects receive standard at SLT at study entry. Subjects who reach Month 12 without discontinuing study treatment are randomized to annual low-energy repeat SLT or as-needed standard energy repeat SLT. There are 2 arms in the first 12 months of the study and 2 arms in Months 13-48.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Trial 1: Initial standard energy SLT (Active Comparator): Standard energy SLT is performed as follows: beginning at 0.8 mJ, energy will be titrated up or down within the first 5-10 spots until champagne bubbles are visualized with every 2nd or 3rd spot. Energy can be titrated throughout the procedure, in response to variations in pigmentation, to ensure the appearance of champagne bubbles with every 2nd or 3rd spot throughout the full 360° treatment. Energy should be increased if no bubbles are seen with 5 consecutive spots and decreased if bubbles are seen with 5 consecutive spots.
  Interventions: Procedure: Standard Energy SLT
- Trial 2: Month 12 Randomization: Annual Low Energy Repeat SLT (Experimental): At month 12, eligible subjects will be randomized to undergo repeat SLT either annually at low energy or as needed at standard energy.
  Low energy SLT will consist of 100 treatment spots delivered at 0.4 mJ per spot throughout the full 360° treatment, with the exception that energy can be reduced to 0.3 mJ if bubbles are seen with 5 consecutive spots and can be increased back to a maximum of 0.4mJ is no bubbles are seen with 5 consecutive spots.
  Interventions: Procedure: Low Energy SLT
- Trial 2: Month 12 Randomization: As-Needed Repeat SLT at Standard Energy (Active Comparator): At month 12, eligible subjects will be randomized to undergo repeat SLT either annually at low energy or as needed at standard energy.
  Standard SLT will be performed as follows: beginning at 0.8 mJ, energy will be titrated up or down within the first 5-10 spots until champagne bubbles are visualized with every 2nd or 3rd spot. Energy can be titrated throughout the procedure, in response to variations in pigmentation, to ensure the appearance of champagne bubbles with every 2nd or 3rd spot throughout the full 360° treatment. Energy should be increased if no bubbles are seen with 5 consecutive spots and decreased if bubbles are seen with 5 consecutive spots.
  Interventions: Procedure: Standard Energy SLT
- Trial 1: Initial Low Energy SLT (Experimental): Note: This arm was discontinued following a planned interim analysis.
  Low energy SLT will consist of 100 treatment spots delivered at 0.4 mJ per spot throughout the full 360° treatment, with the exception that energy can be reduced to 0.3 mJ if bubbles are seen with 5 consecutive spots and can be increased back to a maximum of 0.4mJ if no bubbles are seen with 5 consecutive spots.
  Interventions: Procedure: Low Energy SLT

INTERVENTIONS:
Procedure: Low Energy SLT — SLT performed at low energy
  Arms: Trial 1: Initial Low Energy SLT; Trial 2: Month 12 Randomization: Annual Low Energy Repeat SLT
Procedure: Standard Energy SLT — SLT performed at standard energy
  Arms: Trial 1: Initial standard energy SLT; Trial 2: Month 12 Randomization: As-Needed Repeat SLT at Standard Energy

SUMMARY:
The goal of this study is to understand if SLT performed at low energy is as effective as SLT performed at standard energy, and also to see if repeating SLT at low energy once a year will prevent or delay the need for daily eye drop medications better than waiting for SLT to wear off before repeating it.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older and in good health
2. Each eye with one of the following qualifying diagnoses (diagnoses may differ between eyes):

   1. High-risk ocular hypertension (OHT): IOP > 21 mmHg without glaucomatous optic neuropathy (excavation, diffuse or focal thinning or notching of the neuroretinal rim, visible nerve fiber layer defects, or asymmetry of the vertical cup-to-disc ratio of >0.2 between eyes)
   2. Mild primary open-angle glaucoma: glaucomatous optic neuropathy, visual field mean deviation better than -6.0 dB with no points in the central 5° <15 dB (see figure on next page)
   3. Moderate primary open-angle glaucoma: glaucomatous optic neuropathy, visual field mean deviation equal to or worse than -6.0 dB but no worse than -12.0 dB and no central 5° points <15 dB or mean deviation -12.0 dB or better with 1 central 5° points <15 dB (see figure on next page).
3. Each eye with BCVA 20/200 (UK 6/60) or better

Exclusion Criteria:

1. Use of topical IOP-lowering medications for more than 6 cumulative months at any time in the past 5 years (this is a modification implemented during active enrollment)
2. Any history of IOP-lowering laser (prophylactic iridotomy not included) or surgical procedure
3. Advanced POAG in either eye (worse than moderate POAG as defined above)
4. Glaucoma other than POAG (including pigmentary and pseudoexfoliation glaucoma) in either eye
5. Mean IOP > 35 mmHg at either the screening or baseline visit in either eye
6. Narrow or closed angle (Shaffer Grade 0, 1, or 2) in either eye
7. Contraindications to SLT or any other study intervention
8. Any corneal pathology that would preclude accurate assessment of IOP by Goldmann tonometry in either eye
9. Any intraocular surgical procedure within the past 6 months in either eye
10. Inability to attend all scheduled study visits
11. Pregnant or planning to become pregnant in the next 4 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
12-month survival | 12 months
  Survival of first SLT through Month 12
48-month survival | 48 months
  At Month 12, subjects are randomized to repeat SLT either annually at low energy or PRN at standard energy. The proportion controlled with SLT alone at Month 48 will be compared between groups

SECONDARY OUTCOMES:
Mean IOP | 12 months
  Mean IOP at month 12
Long-term mean IOP | 12, 24, 36, and 48 months
  Mean IOP at each study visit
Incidence of IOP spikes | 0, 12, 24, 36, and 48 months
  IOP spikes > 5 mmHg on day of SLT

CONTACTS AND LOCATIONS:
Overall Officials: Tony Realini, MD, MPH, Study Chair — West Virginia University; Goundappa K Balasubramani, PhD, Principal Investigator — University of Pittsburgh; Stephen Wisniewski, PhD, Principal Investigator — University of Pittsburgh
Locations (29):
- United States (28):
  - Harvard Eye Associates, Laguna Hills, California
  - Doheny Eye Center UCLA, Pasadena, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Mile High Eye Institute, Sheridan, Colorado
  - Clear Vue Laser Eye Center, Lakeworth, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Chicago Arbor Eye Institute, Orland Park, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - Wilmer Eye Institute Johns Hopkins, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Mark Latina, LLC, Reading, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Kresge Eye Institute Wayne State University, Detroit, Michigan
  - New York Eye Surgery Associates, The Bronx, New York
  - University Hospitals Eye Institute, Cleveland, Ohio
  - Cleveland Clinic Cole Eye Institute, Cleveland, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Eye Care Specialists, Kingston, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Ophthalmology Associates, Fort Worth, Texas
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- Ocular Health Centre, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All study data will be de-identified. We will invite other investigators to submit secondary data requests using the data from the study and will work with those investigators to foster additional research studies and manuscripts. The investigators agree to abide by the principles for sharing research resources as described by "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources." All publications based on the study will adhere to the NIH Public Access Policy (Notice NOT-OD-08-033). At the end of the study, all study data will be submitted for permanent archive per the notice of grant award.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study completion
Access Criteria: See above

REFERENCES:
- [Background] Realini T, Gazzard G, Latina M, Kass M. Low-energy Selective Laser Trabeculoplasty Repeated Annually: Rationale for the COAST Trial. J Glaucoma. 2021 Jul 1;30(7):545-551. doi: 10.1097/IJG.0000000000001788. PMID 33428350
- See also: Study website — http://www.COASTtrial.org